CLINICAL TRIAL: NCT07361471
Title: Identification of Genetic, Phenotypic, Clinical, Biological and Histological Factors Differentiating Patients With Ovarian Cancer Who Are Refractory to Platinum-based Therapy From Patients Defined as Long-term Responders to Platinum-based Therapy.
Acronym: ORTRAI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-A01107-42
Record Dates: First submitted 2025-11-28; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; long responder
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: It is a single-centre study with a prospective part (living patients) and a retrospective part (deceased patients) involving data collection via the patient's medical software. A molecular analysis on histological blocks taken at the time of diagnosis will be carried out as part of the study. This analysis may potentially generate new genomic data to classify patients with ovarian cancer. Could result in the incidental discovery of abnormalities, which may eventually modify the management of the patient, notably her monitoring and screening for other pathologies.
  No additional sampling will be carried out as part of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- long-term responders (Experimental): molecular analysis on histological blocks
  Interventions: Genetic: molecular analysis
- refractory patients (Experimental): molecular analysis on histological blocks
  Interventions: Genetic: molecular analysis

INTERVENTIONS:
Genetic: molecular analysis — molecular analysis on histological blocks

SUMMARY:
After having constituted the ORTRAI cohort using the CONSORE database at the Jean PERRIN Center, the objective is to characterize the patients both clinically and biologically, histologically and genomically.

The clinical and biological characterizations will allow us to confirm that our cohort is comparable with data from the literature.

The complement of immunohistochemical and molecular analyses will provide more details on the differences between long-term patients responding to treatment and refractory patients.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, treated at the Jean Perrin Center, suffering from ovarian cancer at any stage and treated with platinum-based chemotherapy in the first line of treatment.
* Corresponding to one of the two groups below:

  * Refractory group: patients progressing in the first therapeutic line of platinum-based chemotherapy.
  * Group of long-term responders: patients who have not progressed 5 years after the end of first-line platinum salt treatment
* Affiliation to a social security scheme
* Patient who signed the genetic consent form

Exclusion Criteria:

* Minor patient
* Pregnant patient
* Patient under guardianship or conservatorship
* Patients who object to the collection of their medical/paramedical data
* Patient for whom the center does not have biological material for genomic analysis (FFPE block)
* Patient under administrative, judicial decision or AME (State Medical Aid)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Molecular anomalies retained after biological interpretation and allowing the differentiation of refractory patients from long-term responder patients. | Through study completion, an average of 1 year
  Refractory patients are defined as any patient progressing through the first therapeutic line of platinum-based chemotherapy.
  Long responders are defined as any patient who has not progressed within 5 years of the end of platinum salt treatment.

SECONDARY OUTCOMES:
Phenotypic criteria differences between refactory patients and long responder patients | Through study completion, an average of 1 year
  Phenotypic criteria will include BMI, personal history and family history
Clinical criteria differences between refactory patients and long responder patients | Through study completion, an average of 1 year
  Clinical criteria will include age at diagnosis, FIGO stage, initial PCI score, CCO score
Biological criteria difference between refactory patients and long responder patients | Through study completion, an average of 1 year
  Biological criteria include CA-125
Histological criteria differences between refactory patient and long responder patients | Through study completion, an average of 1 year
  Histological criteria include histological type, presence of emboli, Ki-67, RO, RP, WT1, PAX8, PD-L1, CD8, p53, HER2

CONTACTS AND LOCATIONS:
Overall Officials: Tressie HERRMANN, MD, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, PUY DE DOME, France

IPD SHARING:
Plan to Share IPD: No